CLINICAL TRIAL: NCT07080333
Title: BLADDER MICROBIOTA AND BLADDER CANCER
Brief Title: MICROBIOTA AND BLADDER CANCER
Acronym: MICROBLADDERK
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 23-API-02; 2025-A01185-44 (Other: IDRCB)
Record Dates: First submitted 2025-07-15; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Bladder (Urothelial, Transitional Cell) Cancer
Keywords: bladder; cancer; microbiota
MeSH Terms: conditions — Neoplasms | interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patient with suspected bladder cancer (Experimental)
  Interventions: Biological: biopsy

INTERVENTIONS:
Biological: biopsy — After verifying the patient's identity, obtaining their informed consent and confirming that there are no immediate contraindications to performing biopsies (haemorrhagic and infectious), the patient will be prepared for RTUV, which will be performed by cystoscopy under anaesthesia in the operating theatre.

SUMMARY:
In France, bladder cancer (BC) is the fourth leading cause of cancer (14,000 new cases per year). It affects older men (>60 years old) and smoking is the main identified risk factor (RF). The persistence of a high sex ratio despite the increase in smoking among women has led to research into other environmental RFs for BC, which may include the microbiota.

Recently, the concept of urinary microbiota in asymptomatic patients has been accepted. Studies on the urinary microbiota have shown dysbiosis associated with certain urogenital pathologies. Thus, similar to certain dysbiosis of the colonic mucosa microbiota associated with CRC, it is possible that certain bacteria or viruses in the bladder tissue microbiota may be involved in bladder carcinogenesis. An epidemiological study conducted by our laboratory showed a prevalence of BC of 14% (7/50) in patients carrying the bacterium Actinotignum schaalii in their urine. While studies have analysed the urinary microbiota of patients with BC, those comparing the microbiota of cancerous bladder tissue with that of healthy tissue in patients with BC remain few in number, involve a limited number of patients, use uncontrolled sample collection, and have all used 16S rDNA-targeted metagenomics methods to study the composition of the microbiota. The authors show a difference in biodiversity between the microbiota of cancerous bladder tissue and that of healthy tissue.

The team hopes to confirm these preliminary results with a multicentre study using a more comprehensive genomic method, global metagenomics. The microbiota of cancerous bladder tissue will be compared with that of healthy bladder tissue in the same patient to highlight any bacterial or viral dysbiosis associated with the cancerous area.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Male
* First RTUV for suspected CV in the presence of macroscopic haematuria or other clinical signs and/or urinary cytology and/or cystoscopy and/or imaging tests suggestive of CV
* Signed informed consent form
* Affiliation with a social security scheme

Exclusion Criteria:

* Antibiotic use within 3 months prior to inclusion
* Current urinary tract infection (urine culture recommended by the AFU prior to RTUV)
* History of surgical treatment of the urinary and genital tracts within the last 6 months prior to inclusion
* History of RTUV
* History of pelvic radiotherapy
* Interstitial cystitis
* Patients with an indwelling urinary catheter
* Vulnerable patients: minors, patients under guardianship or curatorship
* Patients with benign tumours after receipt of the pathological report (inverted papilloma, non-tumour inflammatory lesion)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-10-30 (Estimated)

PRIMARY OUTCOMES:
The biodiversity of the bacterial bladder microbiota by global metagenomics | 36 months
  description of biodiversity of bacterial bladder microbiota

SECONDARY OUTCOMES:
Global biodiversity of viral microbiota by metagenomics | 36 months
  description of global biodiversity of viral microbiota

CONTACTS AND LOCATIONS:
Locations (8):
- France (8):
  - Cannes Hospital, Cannes
  - Marseille university Hospital, Marseille
  - Menton Hospital, Menton
  - Nice University Hospital, Nice
  - Nimes University hospital, Nîmes
  - Paris University Hospital, Paris
  - Rennes University Hospital, Rennes
  - Tours University Hospital, Tours

IPD SHARING:
Plan to Share IPD: No